CLINICAL TRIAL: NCT01844167
Title: The Effect of Noxipoint™ Therapy Versus Physical Therapy With Transcutaneous Electrical Never Stimulation on Chronic Cervical Pain
Brief Title: The Effect of Noxipoint Therapy Versus Physical Therapy With TENS on Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Pain Cure Center, California (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201302023RINB
Record Dates: First submitted 2013-04-22; First posted 2013-05-01 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Cervical Pain
Keywords: noxipoint; physical therapy; cervical pain; trigger point; neck pain; TENS; transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Neck Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical therapy arm (PT) (Active Comparator): * The TENS device used: FDA K071951
  * Patients will be treated with standard physical therapy, including the electrical stimulation. Manual therapy, cold/heat therapy or exercise will be applied at the discretion of the physical therapist for about 60 minutes in each session. Patient education and self-care instructions will be provided. TENS will also be performed in each session for about 30 minutes based on the typical PT guidelines, which will serve both as a part of the standard of care and as a placebo equivalent. It will typically be set at Normal/Modulate mode and 120 Hertz rate.
  Interventions: Procedure: Noxipoint Therapy (NT)
- Noxipoint Therapy arm (NT) (Experimental): Patients will be treated with TENS following Noxipoint Therapy guidelines as highlighted below:
  * The TENS device used: FDA K071951
  * TENS is calibrated to allow for maximum range in the specifications.
  * A pair of electrode pads is placed at the corresponding pair of Noxipoints of the injured muscle/soft tissue, for about 2- 5 minutes during each application.
  * The electrical stimulation is set to induce the C-fiber response based on the feedback of the patient.
  * If the corresponding pain is not eliminated or reduced after a couple of applications on correct Noxipoints, apply an ice pack for about 10-15 minutes on site before and during the next Noxipoint stimulation.
  Interventions: Procedure: Physical therapy(PT)

INTERVENTIONS:
Procedure: Noxipoint Therapy (NT) — • For severe chronic neck pain patients, cervical braces are recommended within the first 2-3 days of each treatment session. The patient has to avoid using the treated tissues/muscles during the "Rest Period": Similar to all other cells, the muscle cell healing or regeneration takes time. Patients are instructed not to use the newly recovered muscle/tissue during the "Rest Period", which is about three days if they are forty or younger, plus about one extra day for every 10 additional years of age. If the patient has extensive injured muscles, take two more days of rest. Ice packs may be used during or soon after the session to prevent Delayed Onset of Muscle Soreness (DOMS) from the TENS stimulation.
  Other Names: Charles Koo's Pain Cure Therapy
  Arms: Physical therapy arm (PT)
Procedure: Physical therapy(PT) — •Placebo effect consideration: TENS is included in both arms to obfuscate the process. Using TENS in the PT arm serves both as a sham-therapy-equivalent to what is used in the NT arm to neutralize placebo bias, and as a meaningful therapeutic remedy. The subject is thus blinded. Placebo effect consideration: TENS is included in both arms to obfuscate the process. Using TENS in the PT arm serves both as a sham-therapy-equivalent to what is used in the NT arm to neutralize placebo bias, and as a meaningful therapeutic remedy. The subject is thus blinded.
  Arms: Noxipoint Therapy arm (NT)

SUMMARY:
Chronic cervical pain is a common problem in rehabilitation clinic, but the treatment is time consuming and the effect unsatisfactory. Noxipoint® Therapy, developed by Dr. Charles C. Koo, is a unique electrical stimulation precisely on corresponding "Noxipoints®" of each injured soft tissue, with specific duration and intensity of TENS that induce C-fiber nerve ending sensation. Each application typically last for 2 to 5 minutes. Based on observations of the clinical application, Noxipoint® Therapy appears to relieve chronic neck and shoulder pain significantly with lasting effect, and effectively improves the range of motion. However, large-scale double-blinded, randomized control study on the therapy is not available yet.

The purpose of this study is to compare the effect of Noxipoint® Therapy and physical therapy (including the current TENS application) on patients with chronic neck pain. This study is a prospective stratified randomized control trial. Eighty subjects with chronic cervical pain will be recruited from the Rehabilitation Department or the Physical Therapy Center of National Taiwan University Hospital (NTUH). The qualified subjects will be stratified and randomly allocated into two arms, 40 persons in each:

1. Physical Therapy group (PT)
2. Noxipoint Therapy group (NT) Subjects in either group will be treated for up to 6 sessions within 3 weeks, about 1.5 hours per session. The treatment will terminate after six sessions or earlier if the patient shows no symptoms.

Subjects will be evaluated before and after the first treatment session and followed up at about 4 weeks, 8 weeks, and 12 weeks after the first treatment.

Outcome measures are (1) the pain scale in the Brief Pain Index, (2) cervical Range of Motion (ROM), (3) Quality of Life (QoL) measured with the Interference of Pain to Life section in the Brief Pain Index (BPI) and (4) ultrasound elastogram. Pain scale, ROM and QoL measures will be taken before and after the first treatment session, and at 4 weeks, 8 weeks and 12 weeks after the first session. Elastogram will be taken before the first treatment, and about four weeks after the first treatment.

Statistics: The effects of PT and NT will be compared based on two-sample hypothesis testing methods. All the estimated P-values are two tailed.

DETAILED DESCRIPTION:
Purpose To compare the effect of Noxipoint™ Therapy and physical therapy on subjects with chronic neck pain.

Background There are many interventions for managing the chronic neck pain. The approaches include physical therapy, medication and local corticoid injection, of which physical therapy (PT) is the most prevalent treatment. Transcutaneous electrical nerve stimulation (TENS) is one of the regular treatments of PT and usually used in chronic neck pain as an adjunct therapy. However, the application of TENS, including the location, duration and intensity of stimulation, is only loosely defined and largely decided by physical therapists and thus vary substantially from one application to another.

In spite of the long history of TENS uses, the results of existing studies, including randomized controlled trials (RCTs), have been inconclusive, with some showing benefits of TENS, and others showing none. Moreover, the studies that cite some positive effect of TENS over placebo also found that the effect does not last in the long run. The only conclusion that could be drawn is that TENS sometimes relieves pain in the short term.

Noxipoint™ Therapy, a particular combination of precise location, intensity and duration of electrical stimulation, invented by Charles Koo, the Co-PI of this protocol, may relieve general muscular-skeletal pain and recover the muscle function permanently. Based on observations of clinical application of Noxipoint Therapy on the neck and the shoulder pain, Noxipoint Therapy showed rapid relief and lasting effect several months after the treatment. However, a large-scale randomized control study is not available yet.

The key point of Noxipoint Therapy is that the location of stimulation is the determining factor of the efficacy of the pain treatment. In addition, the intensity, wave pattern and duration of stimulation also play important roles. The patient's compliance with the instruction to avoid stressing the newly recovered muscle/tissue during the "rest period" is also mandatory.

The purpose of this study is to compare the effect of Noxipoint Therapy and physical therapy on patients with chronic neck pain.

Study design

1. Prospective, patient- and assessor-blinded, stratified, randomized control trial. Stratification factor is the patient-reported primary measure (the pain scale) as described below. Patients will be assigned to two tiers before randomization.
2. Outcome measures: (1) pain scale measured in Brief Pain Index (BPI) from 0 to10 (2) cervical Range of Motion (ROM), (3) Quality of Life (QoL) using BPI Interference of Function, and (4) ultrasound elastogram. The primary outcome is BPI-at-its-Worst. Cervical ROM is used to measure functional restoration, BPI Interference of Functions is used to measure the quality of life, and elastogram is used to evaluate the myofascial condition.

Subject enrollment

1. Subject's inclusion criteria: (1) 20 to 70 years of age, (2) diagnosed as chronic cervical pain syndrome (ICD9: 723.1) (3) having no less than 6 months of the pain history, (4) the pain level >＝ 5 in BPI and (5) with trigger points.
2. Subject's exclusion criteria: (1) cervical spondylosis, (2) local corticoid injection within last two weeks, (3) signs of psychosomatic illness, (4) unwilling to be randomized, (5) pregnant woman.

3.80 subjects will be recruited from the Rehabilitation Department or the Physical Therapy Department of National Taiwan University Hospital (NTUH). After initial evaluation, qualified subjects will be stratified and randomized into the following two arms, about 40 subjects in either arm:

1. Physical Therapy group (PT)
2. Noxipoint Therapy group (NT)

Methods

1. Intervention:

   1. Physical therapy arm (PT):

      * The TENS device used: FDA K071951
      * Patients will be treated with standard physical therapy, including the electrical stimulation. Manual therapy, cold/heat therapy or exercise will be applied at the discretion of the physical therapist for about 60 minutes in each session. Patient education and self-care instructions will be provided. TENS will also be performed in each session for about 30 minutes based on the typical PT guidelines, which will serve both as a part of the standard of care and as a placebo equivalent. It will typically be set at Normal mode and 120 Hertz rate.
   2. Noxipoint Therapy arm (NT): Patients will be treated with electrical stimulation following Noxipoint Therapy guidelines as highlighted below:

      * The TENS device used is the same as in PT. Each is calibrated to allow for maximum range in the specifications.
      * The pair of electrode pads is placed at the skin surface locations of the corresponding pair of Noxipoints of the injured muscle/soft tissue, for about 2- 5 minutes during each application of the electrical stimulation.
      * The electrical stimulation is set to induce the C-fiber response (i.e., dull pain, soreness, or achiness) based on the feedback of the patient during the stimulation.
      * If the corresponding pain is not eliminated or at least reduced after a couple of applications on correct Noxipoints, apply an ice pack for about 10-15 minutes on site before and during the next Noxipoint stimulation to alleviate excessive inflammation.
      * For severe chronic neck pain patients, cervical braces are recommended within the first 2-3 days of each treatment session. The patient has to avoid using the treated tissues/muscles during the "Rest Period": Similar to all other cells, the muscle cell healing or regeneration takes time. Patients are instructed not to use the newly recovered muscle/tissue during the "Rest Period", which is about three days if they are forty or younger, plus about one extra day for every 10 additional years of age. If the patient has extensive injured muscles, take two more days of rest. Ice packs may be used during or soon after the session to prevent Delayed Onset of Muscle Soreness (DOMS) from the TENS stimulation.
      * Placebo effect consideration: TENS is included in both arms to obfuscate the process. Using TENS in the PT arm serves both as a sham-therapy-equivalent to what is used in the NT arm to neutralize placebo bias, and as a meaningful therapeutic remedy. The subject is thus blinded. Placebo effect consideration: TENS is included in both arms to obfuscate the process. Using TENS in the PT arm serves both as a sham-therapy-equivalent to what is used in the NT arm to neutralize placebo bias, and as a meaningful therapeutic remedy. The subject is thus blinded.
   3. Subjects in either group will be treated for up to 6 sessions within 3 weeks, about 1.5 hours per session. The treatment will terminate after six sessions or earlier if the patient shows no symptoms. No additional treatments will be provided after 6 sessions.
2. Evaluation: Pain scale, ROM and QoL will be measured before and after the first treatment and at about 4 weeks and 8 weeks after the first treatment. Pain scale and QoL may be measured before each session, and at 12 weeks (by phone) after the first treatment. Elastogram will be taken before the first treatment and 4 weeks after the first treatment. See attached Time Table at the end.
3. Statistics: The effects of PT and NT will be compared based on two-sample hypothesis testing methods. The significant level is set at 0.05. All the estimated P-values are two tailed. Missing data will be treated using Last Observation Carried Forward (LOCF) method.
4. Safety: Noxipoint Therapy is as safe as any other TENS application, since it is used within the general guidelines of TENS.
5. Patient Data Security Measure: The principle investigators will monitor the data safety with measures, such as keeping the study data separately from its medical data. The mapping table between the subject's identity and a randomly assigned identity will be maintained separately.
6. Compensation: Each subject will be compensated NT$400 for the time/transportation cost; half of which will be for the treatment and the other half for the follow-up. Dropout subjects will be paid pro rata.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 70 years of age
* Diagnosed as chronic cervical pain syndrome (ICD9: 723.1)
* Having no less than 6 months of the pain history
* The pain level >＝ 5 in BPI
* with trigger points.

Exclusion Criteria:

* cervical spondylosis
* local corticoid injection within last two weeks
* signs of psychosomatic illness
* unwilling to be randomized
* pregnant woman

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change of Brief Pain Index (BPI) At Its Worst from baseline to 4 weeks | About 4 weeks after the initial treatment
  BPI At Its Worst will be assessed before the first treatment and followed up at 4 weeks after the start.

SECONDARY OUTCOMES:
Change of the normalized Range of motion(ROM) of the neck from baseline to follow-up at 4 weeks | About 4 weeks after the initial session
Change of BPI Average from baseline to the follow-up at 4 weeks | 4 weeks after the initial treatment
Change of BPI-Right-Now from baseline to the follow-up at 4 weeks | 4 weeks after the initial treatment
Change of BPI-Average from baseline to the follow-up at 8 weeks | 8 weeks after the initial treatment
Change of BPI-Right-Now from baseline to the follow-up at 8 weeks | 8 weeks after the initial treatment
Change of Brief Pain Index (BPI) At Its Worst from baseline to 8 weeks | About 4 weeks after the initial treatment
Change of BPI-Average from baseline to the follow-up at 12 weeks | 12 weeks after the initial treatment
Change of BPI-Right-Now from baseline to the follow-up at 12 weeks | 12 weeks after the initial treatment
Change of BPI At Its Worst from baseline to 12 weeks | 12 weeks after the initial treatment
Change of QoL(Quality of life) from baseline to the follow-up at 4 weeks | 4 weeks after the initial treatment
Change of QoL(Quality of life) from baseline to the follow-up at 8 weeks | 8 weeks after the initial treatment
Change of QoL(Quality of life) from baseline to the follow-up at 12 weeks | 12 weeks after the initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tyng-Guey Wang, MD, Principal Investigator — National Taiwan University; Charles C Koo, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipai, Taiwan